CLINICAL TRIAL: NCT02363894
Title: Directional AthErectomy Followed by a PaclItaxel-Coated BalloN to InhibiT RestenosIs and Maintain Vessel PatEncy: A Pilot Study of Anti-Restenosis Treatment - Two Year Follow-up Extension Study
Brief Title: DEFINITIVE AR Two Year Follow-up Extension Study
Status: Completed | Type: Observational
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-1009
Record Dates: First submitted 2015-02-10; First posted 2015-02-16 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects enrolled in DEFINITIVE AR

SUMMARY:
The purpose of this DEFINITIVE AR Two Year Follow-up Extension Study is to gather data to assess and estimate the long term effect of treating a vessel with plaque excision (PE) in combination with paclitaxel-coated balloon angioplasty (PTX PTA) compared to treatment with PTX PTA alone.

ELIGIBILITY:
Inclusion Criteria:

* Was a subject in DEFINITIVE AR I
* Is able and willing to provide written informated consent prior to study specific data collection.

Exclusion Criteria:

* Withdrew consent in DEFINITIVE AR I.
* Was reported dead during DEFINITIVE AR I.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who participated in DEFINITIVE AR I and completed the 12 month follow-up assessment in DEFINITIVE AR.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Major Adverse Event Rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Thomas Zeller, MD, Principal Investigator — Universitats Herzzentrum Freiburg - Bad Krozingen, Germany; Prof. Gunnar Tepe, MD, Principal Investigator — Klinikum Rosenheim Institut fur Diagnostische und Interventionelle Radiologie - Rosenheim, Germany